CLINICAL TRIAL: NCT00186056
Title: Mifepristone in Refractory Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Hugh Brent Solvason, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 78804
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Mifepristone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mifepristone (Experimental): Patients received mifepristone for 6 days
  Interventions: Drug: Mifepristone
- placebo (Placebo Comparator): Patients received placebo for 6 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Mifepristone — Glucocorticoid antagonist
  Other Names: RU 486
  Arms: Mifepristone
Drug: Placebo Oral Tablet — Inactive placebo tab
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
The purpose of the study is to examine the effectiveness of mifepristone treatment in patients with refractory depression. Refractory depression is defined as clinical depression that is unimproved after treatment with at least 2 different antidepressants of adequate dose and time trial. Mifepristone will augment current medications.

DETAILED DESCRIPTION:
Study Procedures:

This study will be a double-blind placebo-controlled 5-week trial.

Thirty patients with treatment refractory major depression will be studied over a one year period. Patients will be screened for eligibility, no more than two weeks prior to enrollment, which will involve psychiatric interviews (including the SCID-Mini, HAM-D, BPRS, and CGI-S), a physical exam, and blood and urine analyses.

Clinical laboratory assessments include a serum pregnancy test (for all females), comprehensive blood count, comprehensive metabolic panel, lipid panel, fasting insulin, glucose tolerance test, urine toxicology, and electrocardiogram.

If subjects are found to be eligible, they will be asked return within two weeks of their eligibility screening visit to begin the study. Additionally, they will be asked to keep a diary of their sleep pattern for 1 week prior to entering the study and for the entire 5 week duration of the study.

On the day before beginning study medication (Study Day 0), patients will be administered the HAM-D, BPRS, CGI-S, CGI-I and neuropsychological tests, and vitals will be obtained. Patients will also undergo an afternoon blood draw, with a blood sample taken each hour beginning at 1:00PM and ending at 4:00PM, in order to assess baseline cortisol levels. Patients will then be given a 4-day supply of double-blind study medication (either 24 100mg mifepristone tablets or 24 placebo tablets) with instructions to self-administer 6 tablets each morning.

Patients will return on Day 4 to have study staff check on medication adherence, take vitals, and assess any possible adverse events. Patients will then receive an additional 3-day supply of double-blind study medication (either 18 100mg mifepristone tablets or 18 placebo tablets with instructions to orally self-administer 3 tablets each morning.

Patients will return on Day 7 to have study staff check on medication adherence, take vitals, and assess any possible adverse events. Patients will also repeat clinical laboratory assessments (including a serum pregnancy test for all females, comprehensive blood count, comprehensive metabolic panel, lipid panel, fasting insulin, glucose tolerance test, and urinary analysis) and ECG, and repeat the afternoon blood draw from 1:00PM to 4:00PM to assess cortisol levels. They will also be administered the HAM-D, BPRS, CGI-S, and CGI-I.

Patients will return after one week (Day 14) for administration of the HAM-D, BPRS, CGI-S, CGI-I, and assessment of any possible adverse events, and vitals. Patients will also repeat the afternoon blood draw from 1:00PM to 4:00PM to assess cortisol levels.

Patients will also return on Day 28 and Day 35 for administration of the HAM-D, BPRS, CGI-S, CGI-I, and assessment of any possible adverse events, and vitals. All female patients will undergo serum pregnancy testing on Day 35. In addition, all patients will be asked turn in their sleep diary to the research staff and will receive a neuropsychological test on day 35.

During the study, patients will be monitored for adrenal insufficiency and signs of Cushingnoid effects by monitoring blood pressure, pre-treatment (eligibility) and post-treatment (Day 7) metabolic panels (including measures of glucose and potassium), and monitoring of any changes that occur during the study.

Women with child-bearing potential are required to use a double-barrier method to prevent pregnancy during the study and for 30 days after the study. The double-barrier method includes 2 of the following methods of contraception: spermicidal foam, condom diaphragm, or IUD. Women of child-bearing potential are defined as women, 18 years of age or older, who have not been diagnosed by their primary care physician or gynecologist with menopause, and who have an intact uterus. Women not of child-bearing potential are defined as women, 18 years of age or older, who are status post hysterectomy or have been diagnosed by their primary care physician or gynecologist with menopause (as clinically defined by examination and results of FSH/LH blood work).

After the study, subjects will be referred for follow-up care as needed.

Subjects will not be paid for their participation in this protocol.

ELIGIBILITY:
Inclusion Criteria::

* 21-item HAM-D score of 20 or above.
* If currently taking antipsychotic, antidepressant, anticonvulsant, and/or mood-stabilizing medications, must be stable on the medication for at least three weeks prior to entering the study.
* At least 2 failed antidepressant medication trials of adequate dose and duration.
* Between 18 and 75 years of age.
* Not currently pregnant or trying to become pregnant. Exclusion Criteria:-History of schizophrenia or other psychotic disorders.
* Transcranial magnetic stimulation treatment or ECT in the 3 months prior to starting the study.
* History of vagus nerve stimulation treatment.
* No unstable or untreated cardiovascular disease, hypertension, or endocrine disorder.
* Current use of oral contraceptives or any other drug that may result in adverse drug-mifepristone interactions effects (including Amiodarone, Clarithromycin, Erythromycin, Fluconazole, Fluvoxamine, Indinavir, Intraconazole, Ketoconazole, Metronidazole, Miconazole, Nefazodone, Nelfinavir, Norfloxacin, Omeprazole, Quinine, Ritonavir, Saquinavir, Troleandomycin, Zafirlukast, Carbamazepine, Dexamethasone, Ethosuximide, Phenobarbital, Phenytoin, Primidone, Rifabutin, Rifampin, Troglitazone). A 30-day wash-out period for oral contraceptives is required before mifepristone begins.
* Previous allergic reaction to mifepristone or drugs of similar chemical structure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Brent Solvason, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients received placebo for 6 days
  Mifepristone: Glucocorticoid antagonist
Period: Overall Study
Arm/Group | Mifepristone | Placebo
Started | 14 | 17
Completed | 12 | 16
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone | Placebo | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.92 (9.4) | 51.82 (9.6) | 51.43 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 10 | 16
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale
Description: Hamilton Depression Rating Scale. Minimum score of 0 (no depressive symptoms) to maximum of 68 (very severely depressed).
  Outcome Measure is reporting a Change from Baseline in HAMD scores, i.e., scores at Day 35 minus scores at Baseline.
Time Frame: Baseline and Day 35 HAMD scores
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 12 | 16
units on a scale | 18.75 (9.1) | 19.68 (5.5)
Statistical Analysis 1: Comparison: Mifepristone vs Placebo; Test type: Superiority or Other; p < .26, ANOVA; Interaction of HAMD * medication group F(2,26)=1.38, eta sq = .05

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Mifepristone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 0/14 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No